CLINICAL TRIAL: NCT00139399
Title: A Randomised Controlled Trial to Compare Angiographic Patency of Radial Artery Versus Saphenous Vein Used as Free Aorto-coronary Grafts in Coronary Revascularization
Brief Title: Radial Artery Versus Saphenous Vein Patency (RSVP) Study
Acronym: RSVP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: The Royal College of Surgeons of England (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); National Heart Foundation, Australia (Other); Victor Phillip Dahdaleh Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LREC 98-010
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary artery bypass; Coronary arteries; Atherosclerosis; Angiography; Blood flow
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Coronary Artery Bypass; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saphenous vein (Active Comparator): Saphenous vein aortocoronary bypass graft
  Interventions: Procedure: Coronary artery bypass graft (CABG) surgery
- Radial artery (Experimental): Radial artery aortocoronary bypass graft
  Interventions: Procedure: Coronary artery bypass graft (CABG) surgery

INTERVENTIONS:
Procedure: Coronary artery bypass graft (CABG) surgery — Patients were randomized to receive either a radial artery or a long saphenous vein graft to the left circumflex coronary artery territory during CABG surgery

SUMMARY:
The purpose of this study is to determine whether the radial artery (artery in the arm) or saphenous vein (vein in the leg), when used as bypass grafts for coronary artery bypass surgery, have a greater patency rate (degree of opening)at 5 years after surgery.

DETAILED DESCRIPTION:
Arteries differ from veins both in morphology and physiology. Thus the way they behave as in vivo conduits when used in coronary artery bypass grafting is also likely to be different. This may partly explain the predisposition of veins used as coronary conduits to accelerated atherosclerosis in comparison with the internal mammary artery grafts. There are presently few data describing the properties of the radial artery as an in-vivo coronary conduit over the longer-term.

The study will compare angiographic patency of the radial artery or saphenous vein graft anastomosed to the native left circumflex coronary territory at 3 months and 5 years after surgery. A substudy will compare 5-year post-surgery diameter and blood flow of in-vivo radial artery and saphenous vein grafts in response to endothelium-dependent and non-endothelium-dependent stimuli when patients attend for their scheduled follow-up angiogram.

ELIGIBILITY:
Inclusion Criteria:

* on waiting list for clinically-indicated myocardial revascularization surgery
* aged 40-70 years
* significant stenosis (≥70%) in the circumflex territory as identified on preoperative angiograms
* negative Allen's test (defined as the return of palmar circulation within 5 seconds of releasing ulnar artery compression)
* willing to give written informed consent

Exclusion Criteria:

* poor left ventricular (LV) function (LV ejection fraction <25%)
* severe diffuse peripheral vascular disease or bilateral varicose venous disease
* inability to comply with the angiographic follow-up at 3 months or/and 5 years

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 1998-05; Primary Completion 2006-07 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Moat, MS, FRCS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Trust, London, United Kingdom

REFERENCES:
- [Result] Collins P, Webb CM, Chong CF, Moat NE; Radial Artery Versus Saphenous Vein Patency (RSVP) Trial Investigators. Radial artery versus saphenous vein patency randomized trial: five-year angiographic follow-up. Circulation. 2008 Jun 3;117(22):2859-64. doi: 10.1161/CIRCULATIONAHA.107.736215. Epub 2008 May 27. PMID 18506009
- [Result] Chong WC, Collins P, Webb CM, De Souza AC, Pepper JR, Hayward CS, Moat NE. Comparison of flow characteristics and vascular reactivity of radial artery and long saphenous vein grafts [NCT00139399]. J Cardiothorac Surg. 2006 Mar 3;1:4. doi: 10.1186/1749-8090-1-4. PMID 16722590
- [Result] Webb CM, Moat NE, Chong CF, Collins P. Vascular reactivity and flow characteristics of radial artery and long saphenous vein coronary bypass grafts: a 5-year follow-up. Circulation. 2010 Aug 31;122(9):861-7. doi: 10.1161/CIRCULATIONAHA.109.887000. Epub 2010 Aug 16. PMID 20713903

RESULTS

PARTICIPANT FLOW:
Groups:
- Saphenous Vein: Saphenous vein aortocoronary bypass graft
  Patients were randomized to receive a long saphenous vein graft to the left circumflex coronary artery territory during coronary artery bypass graft (CABG) surgery
- Radial Artery: Radial artery aortocoronary bypass graft
  Patients were randomized to receive a radial artery graft to the left circumflex coronary artery territory during coronary artery bypass graft (CABG) surgery
Period: Overall Study
Arm/Group | Saphenous Vein | Radial Artery
Started | 60 | 82
Completed | 44 | 59
Not Completed | 16 | 23

BASELINE CHARACTERISTICS:
Groups:
- Saphenous Vein: Saphenous vein aortocoronary bypass graft
  Patients were randomized to receive a long saphenous vein graft to the left circumflex coronary artery territory during CABG surgery
- Radial Artery: Radial artery aortocoronary bypass graft
  Patients were randomized to receive a radial artery graft to the left circumflex coronary artery territory during CABG surgery
- Total: Total of all reporting groups
Arm/Group | Saphenous Vein | Radial Artery | Total
Number analyzed (Participants) | 60 | 82 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 68 | 109
  >=65 years | 19 | 14 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 58 | 79 | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patency Rates
Description: Angiographic patency rates of radial artery and long saphenous vein grafts at follow-up angiography
Time Frame: 5 years
Population: 103 of the patients randomized at the time of surgery agreed to return for the 5-year follow-up angiogram.
Measure: Count of Participants; unit: Participants
Arm/Group | Saphenous Vein | Radial Artery
Number analyzed (Participants) | 44 | 59
Participants
  Patent graft | 38 | 58
  Occluded graft | 6 | 1

2. Primary Outcome: Mean Diameter of the Study Graft (Saphenous Vein or Radial Artery)
Description: Diameter response of the study vessel (saphenous vein or radial artery graft) to acetylcholine, measured using quantitative coronary angiography from the coronary angiogram.
Time Frame: 5 year follow-up
Population: Intracoronary physiology investigations (diameter and intracoronary Doppler blood flow velocity measurements) were carried out in a subgroup of patients (n=27).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Saphenous Vein | Radial Artery
Number analyzed (Participants) | 12 | 15
mm | 3.18 (0.67) | 2.7 (0.29)

3. Secondary Outcome: Blood Flow Volume
Description: Graft flow response to acetylcholine, calculated from vessel diameter using quantitative coronary angiography, and velocity using an intragraft Doppler wire.
Time Frame: 5 years
Population: 27 of the patients who returned for the 5 year angiogram were eligible for invasive measurement of blood flow.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Saphenous Vein | Radial Artery
Number analyzed (Participants) | 12 | 15
ml/min | 39 (15) | 44 (19)

ADVERSE EVENTS:
Arm/Group | Saphenous Vein | Radial Artery
All-Cause Mortality (participants affected / at risk) | 4/60 | 3/82
Serious Adverse Events (participants affected / at risk) | 11/60 | 13/82
Other Adverse Events (participants affected / at risk) | 0/60 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saphenous Vein (N=60) | Radial Artery (N=82)
Cerebrovascular accident (CVA) (Nervous system disorders) | 2 (2) | 1 (1) — Stroke
Percutaneous coronary intervention (PCI)/angio post surgery (Cardiac disorders) | 7 (7) | 8 (8)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (MI) (Cardiac disorders) | 0 (0) | 2 (2) — Heart attack

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes